CLINICAL TRIAL: NCT06692985
Title: Sentinel Surveillance of Cutaneous Leishmaniasis in Sub-Saharan Africa Based on Non-invasive Molecular Diagnostics: Mapping of Human Cases, Description of Leishamania Species Involved
Brief Title: Epidemiology of Cutaneous Leishmaniasis in Niger, Mali, Togo : Mapping of Clinical Cases, Species, Reservoirs and Vectors of the Disease
Acronym: LEISHAFRICA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Cayenne (Other)
Responsible Party: Sponsor
Other Study IDs: LEISHAFRICA
Record Dates: First submitted 2024-11-06; First posted 2024-11-18 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Cutaneous Leishmaniasis
Keywords: Phylogeny; Sub-Saharian Africa; Mali; Togo; Niger; Sentinel surveillance; Therapeutic
MeSH Terms: conditions — Leishmaniasis, Cutaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Parasitological samples (smear and swabs for PCR)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Single group: Patient of any age with suspicious skin lesions
  Interventions: Other: Clinical and epidemiological data; Other: Parasitological samples; Other: Assessment of clinical course and response to treatment; Other: DLQI questionnaire

INTERVENTIONS:
Other: Clinical and epidemiological data — Collection of clinical and epidemiological data on day 0
Other: Parasitological samples — Parasitological samples : smear for on-site analysis and swabs to be sent to the Cayenne Hospital for PCR at day 0
Other: Assessment of clinical course and response to treatment — Follow-up visit with assessment of clinical course and response to treatment at M6
Other: DLQI questionnaire — DLQI questionnaire at M6

SUMMARY:
Cutaneous leishmaniasis is a neglected tropical disease caused by parasites belonging to the genus Leishmania. This infection can cause skin and sometimes mucous membrane lesions with significant damage. LC has been little studied in sub-Saharan Africa where its incidence is probably underestimated, especially in West Africa. Leishmania major is almost the only isolated species in this region, although recent data suggest the existence of other species, such as L. enrietti. It is said that CL is only present in the arid areas of Africa, but recent outbreaks in wetlands and forests tend to contradict this theory. Due to the lack of availability of the PCR method, the diagnosis of LC in West Africa, especially in Mali, is rarely confirmed. Treatment options are also scarce and their effectiveness is poorly documented. The objectives of this study are to map the occurrence of LC cases with molecular biology confirmation in Niger, Mali and Togo; to determine the different species involved in human cases; evaluate the different treatment options available.

DETAILED DESCRIPTION:
Leishmaniasis is a parasitosis common to humans and animals (anthropozoonosis), caused by flagellated protozoa called Leishmanias, transmitted by the infective bite of the blood-sucking female of a dipteran insect called sandfly. The parasite reservoirs are wild rodents, humans, dogs. Many species of leishmania can infect humans with a multiplicity of clinical pictures that include visceral, localized, diffuse cutaneous forms and mucocutaneous forms.

Cutaneous leishmaniasis (CL) is a neglected tropical disease whose transmission to humans is based on the bite of sandflies previously contaminated on mammalian reservoirs. Worldwide, more than 200,000 new cases are reported annually. While the Americas and the Near or Middle East are the most important areas, sub-Saharan Africa is also concerned. In a systematic review of the literature published in 2018, Sunyoto et al. identified 54 clinical and epidemiological studies on LC in sub-Saharan Africa. Publications were found in 13 of the 48 countries in sub-Saharan Africa. This review highlighted inconsistent case reporting, clear under-publication and data gaps regarding the exact incidence of CL and its transmission factors, particularly in West Africa.

Indeed, cutaneous leishmaniasis is widely described in East Africa, where many studies have been carried out in Ethiopia, Kenya and Sudan. The presence of Leishmania major and Leishmania aethiopica is well documented, and the dynamics of the infection and its risk factors are studied. In West Africa, on the other hand, the data are more fragmented. The disease is historically reported in the "Cutaneous Leishmaniasis Belt", a Sahelian strip of semi-arid zones extending from Senegal to Sudan. WHO nevertheless estimates that the real number of LC contaminations in the sub-region is 5 to 10 times higher than reported.

Thus, no cases were reported between 2015 and 2017 in the sub-region, which is not very credible in view of the dynamics of declarations during the previous or following years. Over the period 2004-2008, only 155 cases per year were reported, across the following countries: Ghana, Mali, Cameroon, Nigeria, Senegal, DRC and Ivory Coast. No data were available for neighbouring countries with similar ecological contexts, such as Niger, Benin, Guinea or Burkina Faso. The latter is probably the country reporting cases on the most regular basis, with between 500 and 1500 cases/year between 1995 and 2015. Nevertheless, no case was reported between 2007 and 2010, which seems difficult to explain scientifically and again testifies to a lack of diagnosis or reporting.

WHO establishes " country profiles " on the epidemiology of LC for each endemic country and designs regional programmes to control the disease. It should be noted that while East African countries such as Kenya or Ethiopia have a well-documented profile, no profile is available for West African countries. In addition, no regional programme has been set up for sub-Saharan Africa, unlike the Americas, South-East Asia, the Eastern Mediterranean or Europe regions. These absences show how neglected this public health problem is in the African region.

Ghana was considered non-endemic to CL until a major outbreak in 2002-2003. More than 2000 cases were then diagnosed, and this after an active screening, following an initial epidemic signal of only about fifteen cases. It is therefore possible that other epidemics, or even a sporadic presence, have remained undetected in some areas of the country. It should be noted that the region of the epidemic (Ho district, Volta region) was bordered by neighbouring Togo, and the testimonies collected in the affected communities suggested an imported pathology. Moreover, it should be noted that this epidemic area in Ghana was located in a forest region, therefore ou tside the LC Belt classically described and the semi-arid areas generally incriminated. This example illustrates the need to explore the epidemiology of LC in areas that are considered non-endemic by their climate.

In a later study carried out in 2015 in 15 villages affected by this epidemic, samples were taken to isolate strains belonging to the Leishmania enriettii complex from three crops. This rarely described species was not generally considered pathogenic to humans. This example illustrates the need for better species diagnosis in some areas where Leishmania major is considered to be the only species involved, although recent data do not support this statement with certainty. The diagnosis of cutaneous leishmaniasis in West Africa is too often based on a simple clinical diagnosis, sometimes supported by a parasitological smear. However, this does not allow the diagnosis of the offending Leishmania species. The lack of molecular biology in isolated areas or populations with limited resources prevents precise knowledge of the species involved.

As for the treatment, it is often inaccessible due to its price or the logistical constraints related to transport. Meglumine antimoniate is the first-line treatment in Senegal but rarely available, while metronidazole is used in Niger. However, its effectiveness has not been strongly demonstrated. In Mali, dermatologists use cryotherapy and thermotherapy, and more rarely meglumine antimoniate. Cyclin-based ointments are also used to treat bacterial superinfection.

Across the subregion, patients are frequently lost to follow-up, due to the high cost of transport for populations in rural areas, which are mainly at risk. The lack of follow-up consultations does not make it possible to reliably assess the proportion of patients who recover spontaneously, those requiring active treatment, the effectiveness of the various treatments offered as well as the possible sequelae (disfiguring scars, etc.) in the absence of active treatment. A prospective cohort with active patient follow-up would provide valuable data to assess whether or not new treatment options are needed.

Overall, it therefore seems relevant to map more precisely the incidence of LC in West Africa, to identify in molecular biology the Leishmania species responsible, to deepen knowledge on the vectors and reservoirs involved and to evaluate the effectiveness and usefulness of current therapeutic options.

ELIGIBILITY:
Inclusion Criteria:

* Clinical suspicion of cutaneous leishmaniasis during a consultation in one of the partner centres (or by the country physicians) = presence of an ulcerative lesion, papules or nodules
* Obtaining informed and voluntary consent

Non inclusion / Exclusion Criteria:

* Objection to the use of their data and/or the taking of the questionnaire
* Refusal to participate
* Withdrawal of participation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The human study population will consist of all subjects of all ages with suspicious skin lesions.
Sampling Method: Non-Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Presence of a positive test (smear or PCR) for Leishmaniasis Cutaneous (LC) | Day 0
  Presence of a positive test (smear or PCR) for Leishmaniasis Cutaneous (LC) at Day 0

SECONDARY OUTCOMES:
Leishmania species | Day 0
  DNA (DesoxyriboNucleic Acid) sequences of Leishmania species identified in PCR at Day 0
Number of participants with therapeutic failure or success | Month 6
  Number of participants with therapeutic failure or success defined as follows:
  * Therapeutic success: re-epithelialization/collapse of all lesions
  * Therapeutic failure: re-epithelialization/collapse of less than 100% or less than 50% of lesions (criteria recommended in international studies according to Olliaro et al. (Plos Negl Trop Dis 2017) Therapeutic failure or success should be assessed at least six weeks according to international recommendations. The follow-up visit may take place between 3 and 6 months after the initial visit.
Presence of scars with impact on quality of life | Month 6
  Presence of scars with impact on quality of life measured by the DLQI (Dermatology Life Quality Index) Dermatology Life Quality Index (DLQI) scores assess quality of life in a wide range of dermatological conditions (non-specific to dermatological conditions).
  It is easy to implement and assesses the impact of the disease on daily activities, including work, social activities and intimate relationships. The scores ranges from 0 to 30 (most impaired quality of life) and correlates well with disease severity :
  No effect: 0 - 1 Low effect: 2 - 5 Moderate effect: 6 - 10 Important effect: 11 - 20 Extremely important effect: 21 - 30

CONTACTS AND LOCATIONS:
Overall Officials: Romain BLAIZOT, MCU-PH, Principal Investigator — Centre Hospitalier de Cayenne (CHC)
Locations (3):
- Faculté de Médecine et d'Odonto-Stomatologie / Université des Sciences, des Techniques et des Technologies de Bamako, Mali, Bamako, Mali, Mali
- Faculté de médecine/Université André Salifou BP806 Zinder NIGER, Zinder, Niger, Niger
- Service de Dermatologie, CHR TSEVIE, Faculté des Sciences de la Santé, Université de Lomé, Lomé, Togo, Togo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Alvar J, Velez ID, Bern C, Herrero M, Desjeux P, Cano J, Jannin J, den Boer M; WHO Leishmaniasis Control Team. Leishmaniasis worldwide and global estimates of its incidence. PLoS One. 2012;7(5):e35671. doi: 10.1371/journal.pone.0035671. Epub 2012 May 31. PMID 22693548
- [Background] Sunyoto T, Verdonck K, El Safi S, Potet J, Picado A, Boelaert M. Uncharted territory of the epidemiological burden of cutaneous leishmaniasis in sub-Saharan Africa-A systematic review. PLoS Negl Trop Dis. 2018 Oct 25;12(10):e0006914. doi: 10.1371/journal.pntd.0006914. eCollection 2018 Oct. PMID 30359376
- [Background] Eshetu B, Mamo H. Cutaneous leishmaniasis in north-central Ethiopia: trend, clinical forms, geographic distribution, and determinants. Trop Med Health. 2020 Jun 3;48:39. doi: 10.1186/s41182-020-00231-w. eCollection 2020. PMID 32518497
- [Background] Tamiru HF, Mashalla YJ, Mohammed R, Tshweneagae GT. Cutaneous leishmaniasis a neglected tropical disease: community knowledge, attitude and practices in an endemic area, Northwest Ethiopia. BMC Infect Dis. 2019 Oct 16;19(1):855. doi: 10.1186/s12879-019-4506-1. PMID 31619180
- [Background] Pareyn M, Van den Bosch E, Girma N, van Houtte N, Van Dongen S, Van der Auwera G, Massebo F, Shibru S, Leirs H. Ecology and seasonality of sandflies and potential reservoirs of cutaneous leishmaniasis in Ochollo, a hotspot in southern Ethiopia. PLoS Negl Trop Dis. 2019 Aug 19;13(8):e0007667. doi: 10.1371/journal.pntd.0007667. eCollection 2019 Aug. PMID 31425506
- [Background] Boakye DA, Wilson M, Kweku M. A review of leishmaniasis in west Africa. Ghana Med J. 2005 Sep;39(3):94-7. PMID 17299551
- [Background] Kweku MA, Odoom S, Puplampu N, Desewu K, Nuako GK, Gyan B, Raczniak G, Kronmann KC, Koram K, Botero S, Boakye D, Akuffo H. An outbreak of suspected cutaneous leishmaniasis in Ghana: lessons learnt and preparation for future outbreaks. Glob Health Action. 2011;4. doi: 10.3402/gha.v4i0.5527. Epub 2011 Jul 13. PMID 21765823
- [Background] Kwakye-Nuako G, Mosore MT, Duplessis C, Bates MD, Puplampu N, Mensah-Attipoe I, Desewu K, Afegbe G, Asmah RH, Jamjoom MB, Ayeh-Kumi PF, Boakye DA, Bates PA. First isolation of a new species of Leishmania responsible for human cutaneous leishmaniasis in Ghana and classification in the Leishmania enriettii complex. Int J Parasitol. 2015 Sep;45(11):679-84. doi: 10.1016/j.ijpara.2015.05.001. Epub 2015 Jun 19. PMID 26099650
- [Background] Diadie S, Diatta BA, Ndiaye M, Seck NB, Diallo S, Niang SO, Dieng MT. Cutaneous leishmaniasis in Senegal: a series of 38 cases at the Aristide Le Dantec University Hospital in Dakar. Med Sante Trop. 2018 Feb 1;28(1):106-108. doi: 10.1684/mst.2017.0722. PMID 29226827
- [Background] Traore B, Oliveira F, Faye O, Dicko A, Coulibaly CA, Sissoko IM, Sibiry S, Sogoba N, Sangare MB, Coulibaly YI, Traore P, Traore SF, Anderson JM, Keita S, Valenzuela JG, Kamhawi S, Doumbia S. Correction: Prevalence of Cutaneous Leishmaniasis in Districts of High and Low Endemicity in Mali. PLoS Negl Trop Dis. 2017 Feb 15;11(2):e0005379. doi: 10.1371/journal.pntd.0005379. eCollection 2017 Feb. PMID 28199331
- [Background] Kone AK, Niare DS, Thera MA, Kayentao K, Djimde A, Delaunay P, Kouriba B, Giudice PD, Izri A, Marty P, Doumbo OK. Epidemiology of the outbreak, vectors and reservoirs of cutaneous leishmaniasis in Mali: A systematic review and meta-analysis. Asian Pac J Trop Med. 2016 Oct;9(10):985-990. doi: 10.1016/j.apjtm.2016.07.025. Epub 2016 Aug 20. PMID 27794393
- [Background] Oliveira F, Doumbia S, Anderson JM, Faye O, Diarra SS, Traore P, Cisse M, Camara G, Tall K, Coulibaly CA, Samake S, Sissoko I, Traore B, Diallo D, Keita S, Fairhurst RM, Valenzuela JG, Kamhawi S. Discrepant prevalence and incidence of Leishmania infection between two neighboring villages in Central Mali based on Leishmanin skin test surveys. PLoS Negl Trop Dis. 2009 Dec 15;3(12):e565. doi: 10.1371/journal.pntd.0000565. PMID 20016847
- [Background] Paz C, Samake S, Anderson JM, Faye O, Traore P, Tall K, Cisse M, Keita S, Valenzuela JG, Doumbia S. Leishmania major, the predominant Leishmania species responsible for cutaneous leishmaniasis in Mali. Am J Trop Med Hyg. 2013 Mar;88(3):583-5. doi: 10.4269/ajtmh.12-0434. Epub 2013 Jan 16. PMID 23324218
- [Background] Coulibaly CA, Traore B, Dicko A, Samake S, Sissoko I, Anderson JM, Valenzuela J, Traore SF, Faye O, Kamhawi S, Oliveira F, Doumbia S. Impact of insecticide-treated bednets and indoor residual spraying in controlling populations of Phlebotomus duboscqi, the vector of Leishmania major in Central Mali. Parasit Vectors. 2018 Jun 14;11(1):345. doi: 10.1186/s13071-018-2909-2. PMID 29898753
- [Background] Berdjane-Brouk Z, Kone AK, Djimde AA, Charrel RN, Ravel C, Delaunay P, del Giudice P, Diarra AZ, Doumbo S, Goita S, Thera MA, Depaquit J, Marty P, Doumbo OK, Izri A. First detection of Leishmania major DNA in Sergentomyia (Spelaeomyia) darlingi from cutaneous leishmaniasis foci in Mali. PLoS One. 2012;7(1):e28266. doi: 10.1371/journal.pone.0028266. Epub 2012 Jan 20. PMID 22276095
- [Background] Anderson JM, Samake S, Jaramillo-Gutierrez G, Sissoko I, Coulibaly CA, Traore B, Soucko C, Guindo B, Diarra D, Fay MP, Lawyer PG, Doumbia S, Valenzuela JG, Kamhawi S. Seasonality and prevalence of Leishmania major infection in Phlebotomus duboscqi Neveu-Lemaire from two neighboring villages in central Mali. PLoS Negl Trop Dis. 2011 May 10;5(5):e1139. doi: 10.1371/journal.pntd.0001139. PMID 21572984
- See also: Chabasse D, Danis M, Guiguen C. Parasitoses et mycoses des régions tempérées et tropicales. Elsevier Masson. 78 p — https://books.google.com/books/about/Parasitoses_et_mycoses.html?id=Y_DQDwAAQBAJ
- See also: Richard M. Leishmanioses. In : HARRISIN Médecine interne. Arnette. Paris; 1995. 896-899 p — https://compagnon.librairiemedicale.com/complement_ouvrage/harrison/